CLINICAL TRIAL: NCT04845347
Title: A Wearable Morning Light Treatment for Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Leslie Swanson, Associate Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00190163; 1R01MH121531-01A1 (NIH)
Record Dates: First submitted 2021-04-09; First posted 2021-04-14 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Post Partum Depression
Keywords: post partum; depression; light therapy
MeSH Terms: conditions — Depression, Postpartum; Depression | interventions — Ultraviolet Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized using the minimization method. The study team will balance assignment to group based on the following baseline characteristics: baseline Structured Interview Guide For The Hamilton Depression Rating Scale (SIGH-SAD) score, maternal age, parity, and infant age.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bright Light Therapy (Experimental)
  Interventions: Device: Bright Light Therapy
- Dim Light Therapy (Sham Comparator)
  Interventions: Device: Dim Light Therapy

INTERVENTIONS:
Device: Bright Light Therapy — Participants will be provided with active, unaltered Re-Timer glasses that will be worn in the morning daily for 60 minutes for 5 weeks on study.
  Other Names: Re-Timer
  Arms: Bright Light Therapy
Device: Dim Light Therapy — Participants on this arm will wear the placebo version of the Re-Timer fitted with neutral density filters. These will be worn in the morning daily for 60 minutes for 5 weeks on study.
  Other Names: Re-Timer- (placebo version)
  Arms: Dim Light Therapy

SUMMARY:
This study will test a consumer health light therapy device (Re-Timer) for women with postpartum depression to better understand how it affects mood and the body clock (also called the circadian clock).

Eligible participants will be enrolled and randomized after baseline assessments. In addition to using the Re-Timer light for 5 weeks participants will complete questionnaires at various timepoints, record sleep information, wear an actigraph watch, and provide saliva samples. Additionally, the sleep of the participants' infants will also be monitored using an ankle-worn device (actigraph) and sleep diary at certain time-points as this may influence the mother's mood/sleep, and in turn affect the results.

The hypotheses regarding the bright light versus the placebo dim light of the study are:

* morning bright light therapy will produce greater improvement from pre- to post-treatment on the Hamilton Rating Scale for Depression
* morning bright light therapy will lengthen the Phase angle difference (PAD) and this will mediate change in depression symptoms.
* morning bright light therapy will produce greater improvements on self-reported depression symptoms, excessive daytime sleepiness, maternal-infant bonding, social functioning, and sleep-related impairment from pre- to post-treatment.

DETAILED DESCRIPTION:
Please note this project added a sub-study (HUM00235787, IRB approved on 7/31/2024) to the main study. However, the sub-study only applies to some of the participants and there are only exploratory outcomes, therefore, this will not affect the main study registration.

ELIGIBILITY:
Inclusion Criteria:

* less or equal (≤) to 26 weeks postpartum
* meet criteria for current major depressive disorder per the Structured Clinical Interview for Diagnostic (SCID) and Statistical Manual of Mental Disorders version 5 (DSM-V)
* not currently receiving treatment for depression (for example, prescription medications or psychotherapy).

Exclusion Criteria:

* Current diagnosis of Posttraumatic stress disorder (PTSD), obsessive compulsive disorder if the onset is outside of the perinatal period, eating disorder, substance abuse or dependence, lifetime history of mania/hypomania or thought disorder per SCID.
* current diagnosis of, or high risk for, sleep-disordered breathing, insomnia disorder, restless leg syndrome, and/or narcolepsy.
* retinal pathology or history of eye surgery
* current use of photosensitizing medications,
* current use of exogenous melatonin or medications that may interfere with the measurement of melatonin (nonsteroidal anti-inflammatory drugs (NSAIDs) if used daily, and beta-blockers)
* medical conditions for which bright light therapy is contraindicated (for example, epilepsy/seizures).
* nightshift work
* currently pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Change in score for the Hamilton Depression Rating Scale (HAM-D total score) | pre-treatment (baseline), post light therapy treatment (approximately week 5)
  Clinician-rated depression symptom severity measure; Hamilton Depression Rating Scale (HAM-D) (17 item version) measures depressive symptoms on a continuous scale. Higher scores indicate worse outcomes. Scores can range from 0 - 52, where 0 means no depression, and 52 is the greatest possible depression. Generally, scores of 8 or higher represent clinical depression.

SECONDARY OUTCOMES:
Change in Phase angle difference | pre-treatment (baseline), post light therapy treatment (approximately week 5)
  Phase angle difference is calculated as the time interval between the time of dim light melatonin onset and the midpoint of sleep.
Change in score for the structured interview guide score the Hamilton Depression Rating Scale-Seasonal Affective Version (SIGH-SAD total score) | pre-treatment (baseline), post light therapy treatment (approximately week 5)
  Clinician-rated depression symptom severity measure; Hamilton Depression Rating Scale-Seasional Affective Version (SIGH-SAD) (29 item version) measures depressive symptoms on a continuous scale. Higher scores indicate worse outcomes. Scores can range from 0 -73, where 0 means no depression, and 73 is the greatest possible depression. Generally scores of 20 or higher represent clinical depression.
Edinburgh Postnatal Depression Scale (EPDS) total score | pre-treatment (baseline), post light therapy treatment (approximately week 5)
  Self-report of depression symptoms. The Edinburgh Postnatal Depression scale is scored from 0 to 30 where 0 is no depression and 30 is most severe depression.
Epworth Sleepiness Scale (ESS) total score | pre-treatment (baseline), post light therapy treatment (approximately week 5)
  Participants complete this 8 item scale and select response from would never doze (0), to high chance of dozing (3). A score of ≥ 10 indicates excessive daytime sleepiness on the ESS.
Patient Reported Outcomes Measurement Information System (PROMIS) - Satisfaction with Participation in Social Roles (SPSR) total score | pre-treatment (baseline), post light therapy treatment (approximately week 5)
  This is 14 questions regarding social roles where participants select items on a 5-point Likert scale (1) to very much (5). The higher the score the more satisfaction.
Patient Reported Outcomes Measurement Information System Sleep-related impairment (SRI) total score | pre-treatment (baseline), post light therapy treatment (approximately week 5)
  This is an 8 question scale regarding sleep impairment where participants select items on a 6-point Likert scale not at all (0) to very much (5). The higher the score the more impairment.
Social functioning as measured by the Postpartum Bonding Questionnaire (PBQ) total score | pre-treatment (baseline), post light therapy treatment (approximately week 5)
  The PBQ is a is a 25 question self-report measure of maternal-infant bonding. Items are scored on a 6-point Likert scale ranging from 0 (always) to 5 (never), sum score ranging from 0 to 125; high = problematic.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Swanson, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-05-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT04845347/ICF_000.pdf